CLINICAL TRIAL: NCT00062478
Title: Phase 2 Treatment of Adults With Primary Malignant Glioma With Karenitecin
Brief Title: Study of Karenitecin (BNP1350) in Patients With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Crown Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTN20405
Record Dates: First submitted 2003-06-06; First posted 2003-06-12 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2019-07

CONDITIONS: Brain Neoplasms; Malignant Neoplasms, Brain; Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — cositecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Karenitecin for intravenous use
  Interventions: Drug: Karenitecin (BNP1350)

INTERVENTIONS:
Drug: Karenitecin (BNP1350) — Karenitecin 1.0 mg/m2 administered as a single 60-minute IV infusion daily for five consecutive days. The cycle is repeated every 21 days until occurrence of progressive disease or unacceptable toxicity.
  Other Names: Karenitecin also referred to as BNP1350

SUMMARY:
The purpose of this study is to evaluate safety and efficacy ofKarenitecin (BNP1350) as a treatment of adults with brain tumors.

ELIGIBILITY:
* Confirmed diagnosis of a newly diagnosed glioblastoma multiforme or recurrent/progressive glioblastoma multiforme, anaplastic astrocytoma, or anaplastic oligodendroglioma.
* Evidence of measurable recurrent or residual primary CNS neoplasm.
* An interval of at least 3 weeks between prior surgical resection or 6 weeks between prior radiotherapy or chemotherapy, and enrollment on this protocol unless there is unequivocal evidence of tumor progression after surgery, radiotherapy, or chemotherapy.
* Hematocrit > 29%, ANC > 1,500, platelets > 125,000
* Serum creatinine < 1.5 mg/dl, BUN < 25 mg/dl, serum SGOT and bilirubin < 1.5 times upper limit of normal
* Negative pregnancy test for female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-10; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Objective Tumor Response Rate | Randomization to end of treatment

SECONDARY OUTCOMES:
Overall Survival | Randomization to date of death due to any cause
Overall Safety | Randomization to end of study participation

CONTACTS AND LOCATIONS:
Locations (1):
- For Information call 210-614-1701 for a site near you, Durham, North Carolina, United States